CLINICAL TRIAL: NCT06679985
Title: A Randomized Phase 2 Study of Casdozokitug in Combination With Toripalimab Plus Bevacizumab in Participants With Unresectable and/or Locally Advanced or Metastatic Hepatocellular Carcinoma
Brief Title: A Trial of Casdozokitug in Combination With Toripalimab Plus Bevacizumab in Participants With Unresectable and/or Locally Advanced or Metastatic Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Coherus Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHS-388-202
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Unresectable Hepatocellular Carcinoma; Locally Advanced Hepatocellular Carcinoma; Metastatic Hepatocellular Carcinoma; Casdozokitug; Toripalimab; Bevacizumab; HCC; Liver Cancer; IL-27; PD-1
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — toripalimab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Casdozokitug Lower Dose + Toripalimab + Bevacizumab (Experimental)
  Interventions: Drug: Casdozokitug; Drug: Toripalimab; Drug: Bevacizumab
- Arm B: Casdozokitug Higher dose + Toripalimab + Bevacizumab (Experimental)
  Interventions: Drug: Casdozokitug; Drug: Toripalimab; Drug: Bevacizumab
- Arm C: Toripalimab + Bevacizumab (Active Comparator)
  Interventions: Drug: Toripalimab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Casdozokitug — Solution for infusion
  Other Names: CHS-388
  Arms: Arm A: Casdozokitug Lower Dose + Toripalimab + Bevacizumab; Arm B: Casdozokitug Higher dose + Toripalimab + Bevacizumab
Drug: Toripalimab — Solution for infusion
Drug: Bevacizumab — Solution for infusion

SUMMARY:
The main goals of this study are to evaluate the safety and efficacy of casdozokitug in combination with toripalimab plus bevacizumab and to define a recommended dose for casdozokitug in combination with toripalimab plus bevacizumab.

ELIGIBILITY:
Key Inclusion Criteria:

* Unresectable locally advanced or metastatic HCC with diagnosis confirmed by histology/cytology or clinically by American Association for the Study of Liver Diseases criteria in cirrhotic participants.
* Disease that is not amenable to curative surgical and/or locoregional therapies or progressive disease (PD) after surgical and/or locoregional therapies.
* ≥ 1 measurable lesion (per RECIST v1.1) that is untreated.

Exclusion Criteria:

* Has received prior systemic therapy for HCC.
* Has previously received an anti-IL-27 antibody (Ab) or anti-IL-27-targeted therapy.
* Has known fibrolamellar HCC histology, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
* Has moderate or severe ascites.
* Has uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently).

Additional protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | From date of first dose to 90 days after date of last dose (Up to approximately 27 months)
Objective Response Rate (ORR) by Investigator Review According to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to approximately 2 years

SECONDARY OUTCOMES:
ORR by Investigator Review According to HCC Modified RECIST (mRECIST) | Up to approximately 2 years
Duration of Response (DoR) by Investigator Review According to RECIST v1.1 | Up to approximately 2 years
DoR by Investigator Review According to HCC mRECIST | Up to approximately 2 years
Progression-free Survival (PFS) by Investigator Review According to RECIST v1.1 | Up to approximately 2 years
PFS by Investigator Review According to HCC mRECIST | Up to approximately 2 years
Disease Control Rate (DCR) by Investigator Review According to RECIST v1.1 | Up to approximately 2 years
DCR by Investigator Review According to HCC mRECIST | Up to approximately 2 years
Overall Survival (OS) | Up to approximately 2 years
Maximum Concentration (Cmax) | Up to approximately 25 months
Minimum Concentration (Cmin) | Up to approximately 25 months
Time to Cmax (Tmax) | Up to approximately 25 months

CONTACTS AND LOCATIONS:
Locations (44):
- United States (25):
  - Mayo Clinic - Scottsdale, Scottsdale, Arizona
  - University of Arizona - Cancer Center, Tucson, Arizona
  - Beverly Hills Cancer Center, Beverly Hills, California
  - City of Hope, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California
  - Cancer & Blood Specialty Clinic, Lakewood, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - The Winship Cancer Institute Emory University, Atlanta, Georgia
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - University of Kansas Cancer Center, Kansas City, Kansas
  - UofL Health Brown Cancer Center, Louisville, Kentucky
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Christus St. Vincent Regional Medical Center, Santa Fe, New Mexico
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina (UNC) - Chapel Hill, Chapel Hill, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University Comprehensive Cancer Center - Arthur G. James Cancer Hospital and Richard J. Solovev Research Institute (OSUCCC - James), Columbus, Ohio
  - University of Pittsburgh Medical Center (UPMC) - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - UW Carbone Cancer Center - Cancer Connect, Madison, Wisconsin
- Australia (5):
  - Royal Brisbane and Women's Hospital, Herston, Brisbane
  - Bankstown-Lidcombe Hospital, Bankstown, New South Wales
  - Monash Health, Melbourne, Victoria
  - St Vincent's Hospital Sydney, Darlinghurst
  - Linear Clinical Research, Nedlands
- Canada (2):
  - Sunnybrook Health Sciences Centre - Bayview Campus, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
- Hong Kong (3):
  - Prince of Wales Hospital, Shatin, New Territories
  - Queen Mary Hospital, Hong Kong, Pok Fu Lam
  - Humanity & Health Clinical Trial Centre, Hong Kong
- Singapore (3):
  - National Cancer Centre Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Curie Oncology, Singapore
- Taiwan (6):
  - China Medical University Hospital, Taichung, Taichung City
  - National Cheng Kung University Hospital, Tainan, Tainan City
  - National Taiwan University Hospital, Tainan, Taipei City
  - Taipei Veterans General Hospital, Taipei, Taipei City
  - Chi Mei Medical Center, Tainan
  - Linkou Chang Gung Memorial Hospital (CGMHLK), Taoyuan

IPD SHARING:
Plan to Share IPD: No